CLINICAL TRIAL: NCT04976387
Title: Assessing Perceived Quality of Care With Differing Pain Management Protocols After Outpatient Otolaryngology Procedures
Brief Title: Post Operative Analgesia and Patient Satisfaction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 52004443
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain; Patient Satisfaction; Analgesia
Keywords: Otolaryngology; Head and Neck surgery; Outpatient surgery; Same day surgery; Post operative pain; Patient satisfaction; Post operative analgesia; NSAID; Acetaminophen; Hydrocodone
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction; Agnosia | interventions — Hydrocodone; Acetaminophen; oxycodone-acetaminophen; Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of three groups prior to surgery. Patients will be prescribed Hydrocodone/acetaminophen, Ibuprofen, and/or Acetaminophen. Patients assigned to treatment Group 1 will take the opioid medication for initial pain control followed by Ibuprofen if pain is not adequately controlled. Group 2 patients will take Ibuprofen for initial pain control followed by the opioid medication if pain is not adequately controlled. Group 3 patients will take Ibuprofen for initial pain control followed by Acetaminophen if pain is not adequately controlled.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers will not be blinded during the process of recruitment of patients due to necessity of prescribing specific medications. Researchers will be blinded during outcome assessment and data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: Hydrocodone/Acetaminophen and Ibuprofen (Experimental): This group will take Hydrocodone/acetaminophen 5mg/325mg every 6 hours as needed for pain control
  If pain is not controlled after 60 minutes then can take Ibuprofen 600mg every 6 hours as needed for additional pain control.
  Interventions: Drug: Hydrocodone/Acetaminophen 5 Mg-325 Mg ORAL TABLET; Drug: Ibuprofen 600 mg
- Group 2: Ibuprofen and Hydrocodone/acetaminophen (Experimental): This group will take Ibuprofen 600mg every 6 hours as needed for pain control
  If pain is not controlled after 60 minutes then can take Hydrocodone/acetaminophen 5mg/325mg every 6 hours as needed for additional pain control.
  Interventions: Drug: Hydrocodone/Acetaminophen 5 Mg-325 Mg ORAL TABLET; Drug: Ibuprofen 600 mg
- Group 3: Ibuprofen and Acetaminophen (Experimental): This group will take Ibuprofen 600mg every 6 hours as needed for pain control
  If pain is not controlled after 60 minutes then can take Acetaminophen 650mg every 6 hours as needed for additional pain control.
  Interventions: Drug: Ibuprofen 600 mg; Drug: Acetaminophen 650 MG

INTERVENTIONS:
Drug: Hydrocodone/Acetaminophen 5 Mg-325 Mg ORAL TABLET — Patients are instructed to take Hydrocodone/acetaminophen 5 mg-325 mg oral tablets every 6 hours as needed for treatment of severe pain
  Other Names: Norco
  Arms: Group 1: Hydrocodone/Acetaminophen and Ibuprofen; Group 2: Ibuprofen and Hydrocodone/acetaminophen
Drug: Ibuprofen 600 mg — Patients will take ibuprofen 600 mg every 6 hours as needed
  Other Names: Advil, Motrin, NSAID
Drug: Acetaminophen 650 MG — Patients will take Tylenol 650mg every 6 hours as needed
  Other Names: Tylenol
  Arms: Group 3: Ibuprofen and Acetaminophen

SUMMARY:
To understand how patients perceive the quality of care they receive when given different post-operative analgesic medications. Specifically the investigators want to assess whether patients who receive non-opioid analgesia following surgery endorse appropriate quality and satisfaction with their care compared to those who receive opioid medication.

DETAILED DESCRIPTION:
It is routine practice to give analgesic medication after any surgical procedure to provide adequate pain control for patients. However with the increase in abuse of opioid prescription medications, physicians have given a new emphasis to different pain regimens that aim to limit the use of opioid medications. The investigator's previous clinical trial demonstrated that for patients undergoing outpatient otolaryngology procedures, not only does Ibuprofen provide equally effective analgesia compared to opioid medication but it can also decrease overall opioid requirement.

In the current proposed study, the investigators wish to build on previous work. The investigators hypothesize that with the addition of Acetaminophen to Ibuprofen, patients undergoing outpatient otolaryngology procedures may not require opioid analgesia at all. While numerous studies corroborate these results, there is little information about patients' satisfaction with their care in light of a shifting emphasis on decreasing opioid prescription. The primary goal of the current study is to better understand patients' perception of care and level of satisfaction when given opioid versus non-opioid postoperative analgesia. If there is conflicting data with regards to patients reporting adequate pain control but poor satisfaction, then perhaps further public health intervention may be necessary to provide additional patient education to help re-establish appropriate and safe patient expectations for postsurgical analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 89 years of age
* Patients undergoing the following outpatient procedures at a LLUHS associated surgical facility:

  * total or partial thyroidectomy
  * parathyroidectomy
  * parotidectomy
  * submandibular gland excision
  * neck mass excision
  * facial mass excision
  * MOHS defect repair
  * excision of cutaneous lesions
  * Other surgeries may qualify and will be assessed on a case by case basis.

Exclusion Criteria:

* Patients under 18 years old or older than 89 years old
* Those allergic to Hydrocodone, Acetaminophen, or NSAIDS
* Patients who are pregnant
* Patients with chronic medical conditions including hepatic/renal disease that precludes their ability to utilize the study medications.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with post operative pain control | First clinic visit after surgery (7 days)
  Patients will be surveyed if they were satisfied with their pain regimen and efficacy of pain control on a scale of 1-5. With 1 being very unsatisfied and 5 being very satisfied.

SECONDARY OUTCOMES:
Efficacy of analgesic regimen and patient attitudes toward treatment they received | First clinic visit after surgery (7 days)
  Patients attitude and overall experience with regards to their pain management will be assessed via the following questions:
  1. How many total days do you estimate that you required medication for your pain?
  2. If you were in a group that received hydrocodone, how many pills do you estimate that you took?
  3. If you were to have another surgery, would you ask your surgeon for a similar pain regimen?
  4. Was this surgery more painful than you anticipated?

CONTACTS AND LOCATIONS:
Overall Officials: Khanh Nguyen, MD, Principal Investigator — Loma Linda University Health System
Locations (1):
- Loma Linda University Health System, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share participants data after this study is finished with other researchers.

REFERENCES:
- [Background] Wilson N, Kariisa M, Seth P, Smith H 4th, Davis NL. Drug and Opioid-Involved Overdose Deaths - United States, 2017-2018. MMWR Morb Mortal Wkly Rep. 2020 Mar 20;69(11):290-297. doi: 10.15585/mmwr.mm6911a4. PMID 32191688
- [Background] Olfson M, Rossen LM, Wall MM, Houry D, Blanco C. Trends in Intentional and Unintentional Opioid Overdose Deaths in the United States, 2000-2017. JAMA. 2019 Dec 17;322(23):2340-2342. doi: 10.1001/jama.2019.16566. PMID 31846008
- [Background] Gomes T, Tadrous M, Mamdani MM, Paterson JM, Juurlink DN. The Burden of Opioid-Related Mortality in the United States. JAMA Netw Open. 2018 Jun 1;1(2):e180217. doi: 10.1001/jamanetworkopen.2018.0217. PMID 30646062
- [Background] Pruitt LCC, Casazza GC, Newberry CI, Cardon R, Ramirez A, Krakovitz PR, Meier JD, Skarda DE. Opioid Prescribing and Use in Ambulatory Otolaryngology. Laryngoscope. 2020 Aug;130(8):1913-1921. doi: 10.1002/lary.28359. Epub 2019 Nov 27. PMID 31774562
- [Background] Dang S, Duffy A, Li JC, Gandee Z, Rana T, Gunville B, Zhan T, Curry J, Luginbuhl A, Cottrill E, Cognetti D. Postoperative opioid-prescribing practices in otolaryngology: A multiphasic study. Laryngoscope. 2020 Mar;130(3):659-665. doi: 10.1002/lary.28101. Epub 2019 Jun 21. PMID 31225905
- [Background] Foghsgaard S, Foghsgaard J, Homoe P. Early post-operative morbidity after superficial parotidectomy: a prospective study concerning pain and resumption of normal activity. Clin Otolaryngol. 2007 Feb;32(1):54-7. doi: 10.1111/j.1365-2273.2007.01315.x. PMID 17298314
- [Background] Song CM, Ji YB, Bang HS, Kim KR, Kim H, Tae K. Postoperative Pain After Robotic Thyroidectomy by a Gasless Unilateral Axillo-Breast or Axillary Approach. Surg Laparosc Endosc Percutan Tech. 2015 Dec;25(6):478-82. doi: 10.1097/SLE.0000000000000204. PMID 26422088
- [Background] Ilyas AM, Miller AJ, Graham JG, Matzon JL. Pain Management After Carpal Tunnel Release Surgery: A Prospective Randomized Double-Blinded Trial Comparing Acetaminophen, Ibuprofen, and Oxycodone. J Hand Surg Am. 2018 Oct;43(10):913-919. doi: 10.1016/j.jhsa.2018.08.011. PMID 30286851
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Wu AW, Walgama ES, Genc E, Ting JY, Illing EA, Shipchandler TZ, Higgins TS. Multicenter study on the effect of nonsteroidal anti-inflammatory drugs on postoperative pain after endoscopic sinus and nasal surgery. Int Forum Allergy Rhinol. 2020 Apr;10(4):489-495. doi: 10.1002/alr.22506. Epub 2019 Dec 13. PMID 31834679
- [Background] Papoian V, Handy KG, Villano AM, Tolentino RA, Hassanein MT, Nosanov LS, Felger EA. Randomized control trial of opioid- versus nonopioid-based analgesia after thyroidectomy. Surgery. 2020 Jun;167(6):957-961. doi: 10.1016/j.surg.2020.01.011. Epub 2020 Feb 29. PMID 32127178
- [Background] Nguyen KK, Liu YF, Chang C, Park JJ, Kim CH, Hondorp B, Vuong C, Xu H, Crawley BK, Simental AA, Church CA, Inman JC. A Randomized Single-Blinded Trial of Ibuprofen- versus Opioid-Based Primary Analgesic Therapy in Outpatient Otolaryngology Surgery. Otolaryngol Head Neck Surg. 2019 May;160(5):839-846. doi: 10.1177/0194599819832528. Epub 2019 Mar 5. PMID 30832548
- [Background] Gostian AO, Loeser J, Tholen C, Wolber P, Otte M, Schwarz D, Heindl LM, Balk M, Gostian M. Postoperative pain after tonsillectomy - the value of standardized analgesic treatment protocols. Auris Nasus Larynx. 2020 Dec;47(6):1009-1017. doi: 10.1016/j.anl.2020.05.011. Epub 2020 Jun 12. PMID 32536501
- [Background] Hallway A, Vu J, Lee J, Palazzolo W, Waljee J, Brummett C, Englesbe M, Howard R. Patient Satisfaction and Pain Control Using an Opioid-Sparing Postoperative Pathway. J Am Coll Surg. 2019 Sep;229(3):316-322. doi: 10.1016/j.jamcollsurg.2019.04.020. Epub 2019 May 30. PMID 31154092